CLINICAL TRIAL: NCT01099293
Title: Correlation Between Cerebrovascular Reactivity and Hepatic Encephalopathy in Patients With Cirrhosis
Brief Title: Cerebrovascular Reactivity in Hepatic Encephalopathy
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Secretaria de Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, M.D. M.Sc, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: GAS-100-09/10-1
Record Dates: First submitted 2010-03-30; First posted 2010-04-06 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; Psychometric Hepatic Encephalopathy Score; Critical Flicker Frequency; Cerebrovascular Reactivity; Endotoxemia; Transcranial Doppler; Liver Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Endotoxemia; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1. Patients with cirrhosis without hepatic encephalopathy.
  2. Patients with cirrhosis and minimal hepatic encephalopathy.
  3. Patients with cirrhosis and hepatic encephalopathy stage 1.
  4. Healthy subjects willing to participate.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cirrhosis, w/o hepatic encephalopathy: Patients with liver cirrhosis without hepatic encephalopathy by clinical (West-Haven), neurophysiological tests (PHES) nor Critical Flicker Frequency evidence.
- Cirrhosis-minimal hepatic encephalopathy: Patients with cirrhosis, without clinical evidence of hepatic encephalopathy (West Haven 0) and with positive tests for both, PHES and CFF.
- Cirrhosis, Hepatic encephalopathy I: Patients with cirrhosis and clinical evidence of hepatic encephalopathy with a West Haven score of I.
- Control: Healthy subjects willing to participate in the study

SUMMARY:
It has been observed that patients with cirrhosis present a generalized state of vasoconstriction as an homeostatic response to splanchnic arteriolar vasodilatation. On progression of the disease, vascular regulation is mismatched, causing altered systemic blood flow and lose in the cerebrovascular reactivity.

The investigators hypothesize that the altered cerebrovascular reactivity induces neurological disturbances related to hepatic encephalopathy and, therefore, the existence of a correlation between cerebrovascular reactivity and the stage of hepatic encephalopathy.

DETAILED DESCRIPTION:
There is no bibliography that evidenciates a correlation between cerebrovascular reactivity and the stage of hepatic encephalopathy. There are however, papers that reveal generalized systemic vasoconstriction in patients with cirrhosis and others that affirm the presence of vascular disregulation and altered reactivity in the Middle Cerebral Artery in cirrhotic patients. In the other hand, there is published data that correlates the neurological manifestations of diseases characterised by altered blood flow and cerebrovascular reactivity with the degree of the vascular disregulation itself, identified by US Doppler. However, there are no studies correlating transcranial US Doppler findings of cerebrovascular reactivity and hepatic encephalopathy in patients with cirrhosis. Giving its importance to the chance of revealing a new way of pathophysiology and therefore, early therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Liver Cirrhosis

Exclusion Criteria:

* Personal history of surgery in the last 4 weeks
* Diagnosis of Diabetes Mellitus, Hypertension, COPD or liver metabolic diseases (Wilson's disease and hemochromatosis)
* Personal history of stroke and/or cancer
* Use of neuropsychiatric drugs
* Neuropsychiatric disorders (Schizophrenia, bipolar disorder, dementia and Attention-deficit hyperactivity disorder)
* Thyroid disorders without replacement therapy
* Hepatic or renal transplant
* Alcoholism with active ingest of alcohol in the last 6 months
* Pregnancy
* Labour turn-overs

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population from which the cohorts will be selected are from a hospital care population.
  Control group will be selected from the health personal by invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Impaired cerebrovascular reactivity identified with transcranial Doppler ultrasonography of the Media Cerebral Artery. | At time of recruitment (first 3 months)
  Recruitment period is planned for the first 3 months of the study, where outcome messures will be evaluated in a single and unique ocassion, at the time of subject enrollment, due to the characteristics of the study (cross-sectional).

SECONDARY OUTCOMES:
Minimal Hepatic encephalopathy identified with psychometric hepatic encephalopathy score (PHES) and Critical Flicker Frequency (CFF). | At time of recruitment (first 3 months)
  Recruitment period is planned for the first 3 months of the study, where outcome messures will be evaluated in a single and unique ocassion, at the time of subject enrollment, due to the characteristics of the study (cross-sectional).
Hepatic encephalopathy stage I identified clinically and PHES and CFF. | At time of recruitment (first 3 motnhs)
  Recruitment period is planned for the first 3 months of the study, where outcome messures will be evaluated in a single and unique ocassion, at the time of subject enrollment, due to the characteristics of the study (cross-sectional).
Blood samples to measure ammonium, , renin-angiotensin-aldosterone system, endotoxemia and Sb100 | At time of recruitment (3 months)
  Recruitment period is planned for the first 3 months of the study, where outcome messures will be evaluated in a single and unique ocassion, at the time of subject enrollment, due to the characteristics of the study (cross-sectional).

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre-Delgadillo, M.D., M.Sc., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencia Medicas de Nutricion Salvador Zubiran, México, State of Mexico, Mexico